CLINICAL TRIAL: NCT04534504
Title: Sleeve Gastrectomy With Uncut Jejunal Bypass (SG-uncut JJB) Verus Sleeve Gastrectomy in Obese Patients, a Prospective Randomized Controlled Study
Brief Title: Sleeve Gastrectomy With Uncut Jejunal Bypass (SG-uncut JJB) Verus Sleeve Gastrectomy in Obese Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhen Jun Wang (Other)
Responsible Party: Sponsor-Investigator, Zhen Jun Wang, Beijing Chao Yang Hospital, Capital Medical University, Beijing Chao Yang Hospital
Organization: Beijing Chao Yang Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SG-uncut JJB 01
Record Dates: First submitted 2020-08-27; First posted 2020-09-01 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Excessive Weight Loss; Total Weight Loss; Sleeve Gastrectomy; Jejunojejunal Bypass; Uncut
Keywords: sleeve gastrectomy; Jejunojejunal bypass; Weight loss; Complication; SG-uncut JJB
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SG-uncut JJB (Experimental): For SG-uncut JJB procedure, the jejunum was not transected, only 200-cm jejunum 20-cm distal to Treiz ligament was measured and side-to-side jejunojejunal anastomosis was made. And the jejunum 3-5cm distal to the anastomosis was ligated with 10# suture.
  Interventions: Procedure: SG-JJB
- SG-JJB (Active Comparator): For SG-JJB procedure, after SG was finished, the jejunum was transected 20-cm distal to Treiz ligament. After that, another 200-cm jejunum was measured and side-to-side jejunojejunal anastomosis was made. The anastomotic and mesenteric defects were closed by hand suture.
  Interventions: Procedure: SG-JJB

INTERVENTIONS:
Procedure: SG-JJB — Base on SG-JJB procedure, the jejunum was not transected, only 200-cm jejunum 20-cm distal to Treiz ligament was measured and side-to-side jejunojejunal anastomosis was made. And the jejunum 3-5cm distal to the anastomosis was ligated with 10# suture.

SUMMARY:
Among various bariatric procedures, sleeve gastrectomy (SG) and Roux-en-Y gastric bypass (RYGB) are the most frequently performed procedures worldwide. Though SG provides similar weight loss effect to RYGB in short-term follow-up, its long-term and very long-term weight loss effect was reported to be inferior to RYGB. Weight regain after SG remains the major concern after 2-year follow-up due to gradual loss of appetite suppression and lack of malabsorption function. SG plus procedures have been developed to strengthen the effect of SG on diabetes control. It has been reported that SG plus jejunojejunal bypass (SG - JJB) offered better weight loss than SG and similar weight loss to RYGB. The present study aims to evaluate the efficacy and safety of sleeve gastrectomy plus uncut jejunojejunal bypass (SG - uncut JJB).

DETAILED DESCRIPTION:
Among various bariatric procedures, sleeve gastrectomy (SG) and Roux-en-Y gastric bypass (RYGB) are the most frequently performed procedures worldwide. Though SG provides similar weight loss effect to RYGB in short-term follow-up, its long-term and very long-term weight loss effect was reported to be inferior to RYGB. Weight regain after SG remains the major concern after 2-year follow-up due to gradual loss of appetite suppression and lack of malabsorption function. SG plus procedures have been developed to strengthen the effect of SG on diabetes control. It has been reported that SG plus jejunojejunal bypass (SG - JJB) offered better weight loss than SG and similar weight loss to RYGB. The present study aims to evaluate the efficacy and safety of sleeve gastrectomy plus uncut jejunojejunal bypass (SG - uncut JJB).

For SG-JJB procedure, after SG was finished, the jejunum was transected 20-cm distal to Treiz ligament. After that, another 200-cm jejunum was measured and side-to-side jejunojejunal anastomosis was made. The anastomotic and mesenteric defects were closed by hand suture.

For SG-uncut JJB procedure, the jejunum was not transected, only 200-cm jejunum 20-cm distal to Treiz ligament was measured and side-to-side jejunojejunal anastomosis was made. And the jejunum 3-5cm distal to the anastomosis was ligated with 10# suture.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 32.5 kg/m2 with or without T2DM;
* 27.5 kg/ m2 < BMI < 32.5 kg/m2 with T2DM but failed conservative treatment and combined with at least two metabolic diseases or comorbidities;
* Duration of T2DM ≤15 years with fasting Cpeptide ≥ 50% of normal lower limit
* Waist circumference: male ≥ 90 cm, female ≥ 85 cm
* Age within 16~65 years old

Exclusion Criteria:

* Pregnancy;
* A history of mental illness and neurological disease;
* The patient refuses surgery;
* Combined with pituitary tumor;
* Long-term use of antidepressant drugs;
* Long-term use of immunosuppressants;
* Situations in which the investigator or other examiner considers from the enrolled study that there are good reasons for nonconformity: if there are potential inconsistencies with the clinical protocol

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-08-26 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
excessive weight loss | 1 year postoperatively
  Percentage of excess weight loss (EWL) at any time postoperative was calculated as the amount of weight loss divided by the amount of excess weight times 100%.
total weight loss | 1 year postoperatively
  total weight loss compared with preoperative weight

SECONDARY OUTCOMES:
Complications | 30 days postoperatively
  Complications within 30 days postoperatively
operating time | during the operation
  time from opeing of the operation to the end of the operation
intraoperative blood loss | during the operation
  blood loss during the operation

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Jun Wang, Study Chair — Beijing Chao Yang Hospital
Locations (1):
- Beijing Chaoyang Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No